CLINICAL TRIAL: NCT03155776
Title: Ultrasound Assessment of Gastric Volume in Infants Undergoing General Anesthesia: Validation Study
Brief Title: Estimation of Preoperative Gastric Volume Using Ultrasound
Acronym: GUS
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Other Study IDs: H 1703-183-843
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GUS_infants: Infants patient undergoing general anesthesia for abdominal surgery
  Interventions: Diagnostic Test: GUS

INTERVENTIONS:
Diagnostic Test: GUS — gastric volume estimation using gastric ultrasound was performed immediately after anesthetic induction, and after aspirating the residual gastric contents using nasogastric tube

SUMMARY:
Aspiration of gastric contents can be a serious anesthetic related complication. Gastric antral sonography prior to anesthesia may have a role in identifying pediatric patients at risk of aspiration. The investigator examined the relationship between sonographic antral area and endoscopically suctioned gastric volumes infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants undergoing general anesthesia with endotracheal intubation were included in this study

Exclusion Criteria:

* a recent (≤1 month) history of oesophageal or gastric surgery, gastrostomy or ileostomy, diaphragmatic hernia, emergent surgery, or a prolonged duration (>5 min) between completion of US assessment and suctioning of gastric contents

Max Age: 1 Year | Sex: All
Age Groups: Child
Study Population: Infants undergoing general anesthesia for abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
gastric antral cross sectional area | immediate after anesthetic induction within 1 minutes.
  ultrasound assessment of gastric antral cross sectional area

CONTACTS AND LOCATIONS:
Locations (1):
- Jin-Tae Kim, Seoul, South Korea

REFERENCES:
- [Derived] Kim EH, Yoon HC, Lee JH, Kim HS, Jang YE, Ji SH, Cho SA, Kim JT. Prediction of gastric fluid volume by ultrasonography in infants undergoing general anaesthesia. Br J Anaesth. 2021 Aug;127(2):275-280. doi: 10.1016/j.bja.2021.03.039. Epub 2021 May 25. PMID 34045064